CLINICAL TRIAL: NCT01678248
Title: The Effectiveness of Intravitreal Avastin Injection for CRVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0048-12-ZIV
Record Dates: First submitted 2012-08-29; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
to determine the effectivness of intravitreal avastin injection on visual acuity on people that suffer from central retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years old
* suffer from CRVO
* maximal visual acuity 6/15

Exclusion Criteria:

* VA of LP
* retinal disease other than CRVO
* incomplete medical record
* follow up less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who suffer from CRVO and were injected by bevazicumab intravitrealy
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel